CLINICAL TRIAL: NCT04467606
Title: Institutional Review Board Chang Gung Medical Foundation
Brief Title: Motivational Interview Based Discharge Planning for Patients With Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chin yenfan, Assistant Research Fellow, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201901813B0
Record Dates: First submitted 2020-07-04; First posted 2020-07-13 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Diabetic Foot Ulcer
Keywords: Foot ulcer, motivational interviewing, discharge planning
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to either the experimental or the comparison group.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: This study adopted a single blind study design. The research assistants who do not know the research object group perform pre- and post-test data collection, including interviews, medical record data collection and foot evaluation. Due to the different intervention measures received by the experimental group and the control group, we specifically advise the research subjects not to disclose the status of the intervention measures to the research assistant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will receive a discharge planning which use the strategy of motivational interviewing.
  Interventions: Behavioral: a discharge planning using the strategy of motivational interviewing
- Control (No Intervention): Participants will receive routine care of the research setting only. The counseling will be provided if participants request.

INTERVENTIONS:
Behavioral: a discharge planning using the strategy of motivational interviewing — The experimental group will receive a discharge planning which use the strategy of motivational interviewing. The discharge planning will be provided individually at the following time points: before discharge, on post-discharge days 3, 7, 14, 21, 28, and then each month till one year.
  Arms: Experimental

SUMMARY:
To evaluate the effectiveness of a discharge planning using the strategy of motivational interviewing among patients with diabetic foot ulcers

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of a discharge planning using the strategy of motivational interviewing among patients with diabetic foot ulcers.

A randomized controlled trial design will be used. From August 2020 to July 2022, 132 patients hospitalized for diabetic foot ulcers will be recruited. They will be randomly assigned to either the experimental or the comparison group in the first year, and then they will be followed by one year. The control group will receive routine care; the experimental group will receive a discharge planning which use the strategy of motivational interviewing. The discharge planning will be provided individually at the following time points: before discharge, on post-discharge days 3, 7, 14, 21, 28, and then each month till one year. Outcome measures include diabetic foot ulcer self-care behaviors and self-efficacy, foot skin conditions, glycemic control (measured by HbA1C), the infection rate of foot, and the readmission rate. Data will be collected at baseline and at 1, 3, 6, and 12 months after discharge.

The generalized estimating equation (GEE) will be used to evaluate the effect of the intervention on the diabetic foot ulcer self-care behaviors and self-efficacy, foot skin conditions, and the effect on glycated hemoglobin value reduction. The log-rank test will be used to compare the infection rate of foot, and the readmission rate between two groups.

ELIGIBILITY:
Inclusion criteria DFU inpatient Could communicate with Mandarin or Taiwanese HbA1C value higher or equal to 7.5 % Wagner stage 1 or 2 foot ulcer. Exclusion criteria Cognitive impairment Communication problems Affected foot has been amputated Autoimmune disease Be unable to perform daily self-care activity Be cared by foreigner and no other family members live together Plan to move to a long-term care facility Unwilling to visit the outpatient clinic at the research setting C-reactive protein values are higher than 15 mg/dL

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of foot infection and readmission for foot ulcer | 5 minutes
  Foot assessment and the review of medical record

SECONDARY OUTCOMES:
Glycemic control | 1 minutes
  Review the Glycated hemoglobin value on the medical record
Foot skin conditions | 1 minutes
  Foot assessment
Knowledge regarding warning signs of diabetic foot ulcer | 5 minutes
  The WS-DFUD-KQ comprises of 12 items. Three of the 12 items are negatively worded and state as misconceptions regarding warning signs of diabetic foot ulcer deterioration (i.e. item 8, 9, 10). The response choices include "yes," "no," and "uncertain." Each item with the correct answer obtains a score of 1, after which the scores are summed to obtain a total score. The higher scores represent better knowledge. The total WS-DFUD-KQ score ranges 0-12.
  The content validity index of each of the 12 items was above 0.8. The item difficulty of the 12 items of the WS-DFUD-KQ ranged from 0.54 to 0.87, and the item discrimination index D values ranged from 0.42 to 0.83. The KR-20 of the WS-DFUD-KQ was 0.82. The Spearman's rho coefficient for test-retest reliability over a two-week period was 0.75.
Diabetes Foot Self-Care Behavior | 3 Minutes
  The Diabetes Foot Self-Care Behavior Scale (DFSBS) contains 7 items. The scale has two parts: In the first part, the responses are rated on the number of days patients performed a certain behavior over the course of one week. In the second part, the responses are rated by the frequency with which patients performed a certain behavior in general, from never (1) to always (5). When the score of the total scale is calculated, the number of days for each foot-care measure in the first part is categorized across 5 groups (0 days, 1-2 days, 3-4 days, 5-6 days, and 7 days). Thus, all items on the scale are rated on a 5-point Likert-type scale with the higher scores represented better foot self-care behaviors. The total DFSBS score ranges 7-35.
Self-care behaviors of diabetes | 4 Minutes
  The Chinese version of summary of diabetes self-care activity questionnaire (C-SDSCA) is a short self-reported questionnaire of diabetes self-management across five components of diabetes regimen a person with diabetes should practice in order to stay well ( i. e. diet, exercise, blood sugar testing, foot care and attention to smoking). The number of days for each diabetes self-management behavior is measured. The higher scores represented better self-care behaviors of diabetes. The total C-SDSCA score ranges 11-77.
Diabetes-related Foot Ulcer Self-Management Behavior | 9 Minutes
  The Diabetes-related Foot Ulcer Self-Management Behavior Scale (DFUSMBS) measures behaviors that patients use to manage their diabetes-related foot ulcers to promote wound healing and to prevent the deterioration of their wounds, including timely treatment seeking and management, wound management, and self-management of diabetes. The 18-item scale includes three reverse-scored items (Item 1, 2, 11) and uses a 5-point Likert scale (1 = never, 2 = seldom, 3 = sometimes, 4 = frequently, and 5 = always). The higher scores represent better diabetes-related foot ulcer self-management behaviors. The total DFUSMBS score ranges 18-90.
Diabetes management self-efficacy | 10 Minutes
  The Chinese version of the Diabetes Management Self-Efficacy Scale (C-DMSES) is a self-administered scale containing 20 items. It assesses the extent to which respondents are confident that they could manage their blood sugar, diet, and level of exercise. Responses are rated on a 10-point Likert-style from not at all (1) to certainly can do (10). The responses are summed to become a total score for "self-efficacy". Possible scores range from 0 to 200 points. The tool had acceptable reliability and validity in a Taiwanese population.
Self-efficacy regarding diabetes foot self-care | 1 Minute
  Two items will be used to measure the self-efficacy regarding diabetes foot self-care of participants. They are "I have confidence to check my feet (including the bottom of my feet and between the toes) daily, either by myself or to ask for someone's help.", and "I have confidence to apply moisturizing lotion to my feet by myself or asking for someone's help, If my skin is dry". Responses are rated on a 10-point Likert-style scale according the degree of confidence.
Self-efficacy regarding diabetes-related foot ulcer self-management | 5 Minutes
  The 16-item diabetes-related foot ulcer self-management self-efficacy scale will be used to measure the confidence in delivering diabetic foot ulcer self-management behavior, and management of diabetic foot ulcer. Responses are rated on a 10-point Likert-style from not at all (1) to certainly can do (10). The higher score indicates better self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Fan Chin, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

REFERENCES:
- [Derived] Chin YF, Yeh JT, Yu HY, Hsu BR, Lin YJ. A discharge planning program to prevent infection among patients with diabetic foot ulcers in Taiwan: A randomized controlled trial study. J Tissue Viability. 2025 Aug;34(3):100901. doi: 10.1016/j.jtv.2025.100901. Epub 2025 Apr 10. PMID 40280029